CLINICAL TRIAL: NCT01752660
Title: Endurance Training in Severely Disabled Patients With MS - a Feasibility Study
Brief Title: Exercise in Severely Disabled Patients With MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Danish MS Society (Unknown); Danish MS Hospitals, Haslev and Ry (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UAarhus100
Record Dates: First submitted 2012-11-12; First posted 2012-12-19 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Sclerosis
Keywords: Exercise therapy; Aerobic training; Endurance training
MeSH Terms: conditions — Multiple Sclerosis | interventions — Endurance Training; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endurance training (Experimental): Standard care during a 4 week inpatient stay at a Danish multiple sclerosis rehabilitation center added 3 weekly sessions of endurance training for the upper extremity.
  Interventions: Behavioral: Endurance training; Behavioral: Standard care
- Standard care (Active Comparator): Standard care during a 4 week inpatient stay at a Danish multiple sclerosis rehabilitation center
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Endurance training — Standard care during a 4 week inpatient stay at a Danish multiple sclerosis rehabilitation center added 3 weekly sessions of endurance training for the upper extremity.
  Arms: Endurance training
Behavioral: Standard care — Standard care during a 4 week inpatient stay at a Danish multiple sclerosis rehabilitation center.

SUMMARY:
In the last decade physical exercise has become an accepted and integrated part of rehabilitation in patients with multiple sclerosis (MS). However, no studies have evaluated whether the most severely disabled patients can tolerate and benefit from exercise therapy. The purpose of this study is therefore to evaluate the feasibility of endurance training in severely disabled patients with MS.

DETAILED DESCRIPTION:
For many years, patients with multiple sclerosis (MS) have been advised not to participate in physical exercise. This advice was given in part because some patients were reported to experience symptom instability during exercise as a consequence of increased body temperature. A further argument was that avoiding exercise would preserve energy and thereby result in less fatigue, leaving more energy for activities of daily living. During the last decade, it has been more common to recommend exercise for MS patients, because of its recently proven beneficial effects in these patients.

Resistance- and endurance training constitutes the two extremes of basic physical exercise. To gain insight into the effects of exercise it therefore makes sense to understand the extremes. In mild to moderately impaired MS patients endurance training is well tolerated and providing beneficial effects. However, this exercise modality has not yet been tested in severely disabled patients, and it is therefore unclear if endurance training is feasible and beneficial in these patients. The investigators have, therefore, designed a feasibility study evaluating the effects of 4 weeks of endurance training in severely disabled MS patients (Expanded Disability Status Scale score > 6).

Patients are inpatients at one of the national MS hospitals and endurance training is added to the usual care, and compared to usual care only (control group). Exercise frequency is 3 times per week, and intensity is controlled by HR measurements during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  ->18 years
* Primary progressive or secondary progressive MS according to the McDonald criteria
* 6.5 ≤ EDSS ≤ 8.0 and pyramidal score between 1 and 4
* Maximal walking distance ≤ 10m

Exclusion Criteria:

* Patients are excluded if they:
* have dementia,alcoholism, or pacemaker treatment
* any serious medical comorbidities
* are pregnant
* have done systematic endurance training (>1day/week) within the last 3 months.
* complete less than 80% of the planned training sessions
* medical conditions that exclude performance of a maximal endurance test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Exercise compliance | Exercise compliance is registered immediatly after all planned exercise sessions during the 4 week intervention
  Compliance to exercise is registered and serve as the primary outcome.
Drop out rate | Number of participants who drop out is registered at the post measurement just after the intervention.

SECONDARY OUTCOMES:
Peak oxygen consumption | 1-2 day before the intervention and 1-2days after the 4 week intervention peak oxygen is measured
  Measurement of peak oxygen consumption during a ramp protocol on armergometer.
Box and Block test | 1-2 day before the intervention and 1-2days after the 4 week intervention the box and block test is performed
Sit to stand test | 1-2 day before the intervention and 1-2days after the 4 week intervention the sit to stand test is performed
Handgrip test | 1-2 day before the intervention and 1-2days after the 4 week intervention the handgrip test is performed
Wheel-chair test | 1-2 day before the intervention and 1-2days after the 4 week intervention the wheel-chair test is performed

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Dalgas, PhD, Principal Investigator — Dep. Public Health, Aarhus University
Locations (1):
- MS Hospital in Ry, Ry, Jylland, Denmark

REFERENCES:
- [Derived] Skjerbaek AG, Naesby M, Lutzen K, Moller AB, Jensen E, Lamers I, Stenager E, Dalgas U. Endurance training is feasible in severely disabled patients with progressive multiple sclerosis. Mult Scler. 2014 Apr;20(5):627-30. doi: 10.1177/1352458513505351. Epub 2013 Sep 20. PMID 24057428